CLINICAL TRIAL: NCT00391573
Title: Polyglactin Sutures Versus Nylon Sutures for Suturing of Conjunctival Autograft in Pterygium Surgery: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KC/KE-05-0008; HARECCTR0500063
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

INTERVENTIONS:
Procedure: Polyglactin sutures for suturing of conjunctival autograft in pterygium surgery
Procedure: Nylon sutures for suturing of conjunctival autograft in pterygium surgery

SUMMARY:
To compare the use of polyglactin sutures versus nylon sutures for conjunctival autograft suturing in pterygium surgery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included patients with primary nasal pterygium, aged 18 years or older, and able to cooperate surgery under local anaesthesia.

Exclusion Criteria:

* Patients with recurrent pterygium, scarred superior conjunctiva, previous surgery involving the superior bulbar conjunctiva, history of glaucoma, and cicatricial ocular surface disease were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2005-03; Study Completion 2005-06

PRIMARY OUTCOMES:
The difference in VAS score between the two groups

SECONDARY OUTCOMES:
Graft hyperemia, oedema and tarsal conjunctival papillary hypertrophy
Surgical complications
Pterygium recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Wong, Dr, Principal Investigator — Hong Kong Eye Hospital
Locations (1):
- Hong Kong Eye Hospital, Hong Kong, China